CLINICAL TRIAL: NCT02068638
Title: Exercise-related Fuel Metabolism and Glucose Stability in Individuals With Type 1 Diabetes Mellitus
Brief Title: Impact of Physical Activity on Blood Glucose Stability and Energy Stores in Individuals With Type 1 Diabetes
Acronym: CARBEX1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); University of Lausanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 001/14; 320030_149321/1 (Other: Swiss National Science Foundation (SNF)); 191/10 (Other: Ethics Committee (approval of measurements for healthy controls))
Record Dates: First submitted 2014-02-18; First posted 2014-02-21 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes Mellitus; Exercise; Hypoglycemia; Carbohydrate Metabolism
Keywords: exercise; isotope labeling, stable; spectroscopy, magnetic resonance; monitoring, home blood glucose; hormones
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IHE first, CONT second, CSII and MDI therapy (Experimental): IHE: intermittent high intensity exercise: integration of 10 s maximal sprints every 10 minutes in a continuous low to moderate intensity exercise of 90 minutes CONT (occurring after a washout period of 2-8 weeks): continuous moderate intensity exercise of 90 minutes
  Interventions: Procedure: IHE first, CONT second
- CONT first, IHE second,CSII and MDI therapy (Experimental): CONT: continuous moderate intensity exercise of 90 minutes. IHE (occurring after a washout period of 2-8 weeks): intermittent high intensity exercise: integration of 10 s maximal sprints every 10 minutes in a continuous low to moderate intensity exercise of 90 minutes
  Interventions: Procedure: CONT first, IHE second
- GLU first, GLUFRU second, CSII and MDI therapy (Experimental): GLU: ingestion of a 6% carbohydrate solution (consisting of 100 g glucose dissolved in 1000 ml tap water) over a continuous moderate exercise of 90 minutes. GLU FRU (occurring after a washout period of 2-8 weeks): ingestion of a 20% carbohydrate solution (consisting of 100 g glucose + 100 g fructose dissolved in 1000 ml tap water) over a continuous moderate exercise of 90 minutes. CSII = continuous subcutaneous insulin infusion. MDI=multiple daily injections.
  Interventions: Procedure: GLU first, GLU-FRU second
- GLU-FRU first, GLU second, CSII therapy (Experimental): GLU-FRU : ingestion of a 20% carbohydrate solution (consisting of 100 g glucose + 100 g fructose dissolved in 1000 ml tap water) over a continuous moderate exercise of 90 minutes. GLU (occurring after a washout period of 2-8 weeks): ingestion of a 10% carbohydrate solution (consisting of 100 g glucose dissolved in 1000 ml tap water) over a continuous moderate exercise of 90 minutes. CSII = continuous subcutaneous insulin infusion. MDI=multiple daily injections.
  Interventions: Procedure: GLU-FRU first, GLU second

INTERVENTIONS:
Procedure: IHE first, CONT second — IHE: intermittent high intensity exercise: integration of 10 s maximal sprints every 10 minutes in a continuous low to moderate intensity exercise of 90 minutes. CONT (occurring after a washout period of 2-8 weeks): continuous moderate intensity exercise of 90 minutes
  Arms: IHE first, CONT second, CSII and MDI therapy
Procedure: CONT first, IHE second — CONT: continuous moderate intensity exercise of 90 minutes. IHE (occurring after a washout period of 2-8 weeks): intermittent high intensity exercise: integration of 10 s maximal sprints every 10 minutes in a continuous low to moderate intensity exercise of 90 minutes
  Arms: CONT first, IHE second,CSII and MDI therapy
Procedure: GLU first, GLU-FRU second — : ingestion of a 6% carbohydrate solution (consisting of 90 g glucose dissolved in 1500 ml tap water) over a continuous moderate exercise of 90 minutes. GLU FRU (occurring after a washout period of 2-8 weeks): ingestion of a 12% carbohydrate solution (consisting of 90 g glucose + 90 g fructose dissolved in 1500 ml tap water) over a continuous moderate exercise of 90 minutes
  Arms: GLU first, GLUFRU second, CSII and MDI therapy
Procedure: GLU-FRU first, GLU second — GLU-FRU : ingestion of a 12% carbohydrate solution (consisting of 90 g glucose + 90 g fructose dissolved in 1500 ml tap water) over a continuous moderate exercise of 90 minutes. GLU (occurring after a washout period of 2-8 weeks): : ingestion of a 6% carbohydrate solution (consisting of 90 g glucose dissolved in 1500 ml tap water) over a continuous moderate exercise of 90 minutes.
  Arms: GLU-FRU first, GLU second, CSII therapy

SUMMARY:
Whereas physical activity clearly results in improvements in glycemic control in type 2 diabetes, in individuals with type 1 diabetes (T1DM) the impact of exercise on blood sugar control is more complex. In type 1 diabetes T1DM the inability to reduce exogenous insulin levels during exercise is a key factor that contributes to an increased risk of exercise-induced hypoglycemia. Since rapid adaptation of insulin dosage may be especially difficult in patients on a multiple daily injection regimen, alternative strategies are required to improve exercise-associated glucose stability. There is increasing evidence that the combination of steady state continuous low to moderate intensity exercise with short bursts of high intensity exertion (eg in the form of sprints) is an effective, well tolerated, novel strategy to prevent exercise-related hypoglycemia. A further promising option to stabilize blood sugar levels during and after exercise may be the ingestion of fructose in addition to glucose in form of a sport drink.

DETAILED DESCRIPTION:
Background

Regular physical activity enhances insulin sensitivity in both healthy subjects and patients with diabetes mellitus. However, while the effects of physical activity on glucose control are undoubtedly beneficial in patients with type 2 diabetes, exercise can cause major disturbances in blood glucose levels in type 1 diabetic individuals. Hypoglycemia is a common complication in patients with T1DM engaging in endurance activities such as running and cycling. So far there are limited strategies suggested to improve exercise-related blood sugar self-management. Current recommendations focus on variation in timing and dosage of insulin administration and adjustments in carbohydrate intake. Since rapid adaptation of insulin dosage may be difficult, alternative strategies to improve exercise-related glucose stability are required. Increasing evidence suggests that intermittent high intensity exercise (IHE), by triggering a counterregulatory hormone response, may counter-balance the risk of exercise-associated hypoglycemia. However, previous studies investigating IHE in T1DM were limited by heterogeneous study populations, comparably short exercise protocols, and deficits in standardization procedures. In addition, a comprehensive assessment of the underlying fuel metabolism has not been performed so far. As a consequence, the results remain controversial and their interpretation as well as applicability are restricted.

A further alternative strategy to maintain stable glycemia during exercise may be deduced from recent studies in non-diabetic individuals suggesting that the combined ingestion of fructose and glucose during exercise provides the liver with an increased amount of gluconeogenic precursors, thereby reducing consumption of endogenous glycogen stores.Moreover, conversion of fructose into glucose and lactate may provide constant and efficient fuel for working muscles. However, studies assessing the impact of fructose ingestion during exercise in patients with T1DM have not been performed so far.

Objective

The investigators aim to assess the impact of two novel non-pharmaceutical and easily feasible approaches on exercise-related blood glucose stability and its underlying exercise-related fuel metabolism in patients with T1DM.

Substudy A will assess the influence on exercise-related glycemia and fuel metabolism of an IHE protocol compared to an iso-energetic continuous exercise (CONT). It will be investigated whether individuals reach more stable blood glucose levels when engaging in IHE compared to CONT.

Substudy B will investigate whether fueling the patients with a mixed oral 1:1 glucose-fructose carbohydrate solution will maintain glucose values within a more stable range when compared to carbohydrate supplementation by glucose alone.

Methods

Blood glucose levels, counterregulatory hormones, metabolites such as lactate and free fatty acids as well as inflammatory biomarkers will be assessed by regular blood samplings. By means of oral and intravenously given stable isotopes (U-13 C glucose and 2H glucose) exercise-related glucose kinetics will be investigated. Exercise-induced glycogen consumption will be measured using magnetic resonance spectroscopy technology. Late glycemic excursions will be recorded by continuous glucose monitoring systems.

In order to validate 13C magnetic resonance spectroscopy (MRS) measurement of hepatic and myocellular glycogen content a pre-study involving 10 patients and an equal number of matched healthy controls will be performed (validation and reproducibility study).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18 to 35 years
* Diabetes mellitus duration for at least 5 years
* No change in insulin regimen for at least 3 months prior to the study
* Under acceptable to good metabolic control
* Normal insulin sensitivity
* Regular physical activity
* BMI in the range of 18-25 kg/m2
* Written informed consent

Exclusion Criteria

* Diabetes-related complications (macro and microvascular)
* Anemia (hemoglobin concentration <130g/l)
* Abnormal thyroid function
* Dyslipidemia
* Major depression, psychosis and other severe personality disorders, claustrophobia
* Active neoplasia
* Contraindications to exposure to a 3 T magnetic field
* Abnormal liver or renal function
* Smoking, drug abuse, or daily alcohol consumption >60g
* Participation in another study
* Medication other than insulin

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Amount of exogenous glucose required to maintain glycemia within a range between 7-10mM | 30 minutes (last 30 minutes of 90 min exercise period)

SECONDARY OUTCOMES:
Exercise - related glycogen consumption | 90 minutes
Glucose kinetics | 180 minutes
  Rate of glucose appearance and disappearance
Counterregulatory hormones, metabolites, and inflammatory response | 300 minutes
Spiroergometric parameters | 180 minutes
  CO2 and O2 production, RER
Pre- and post-exercise glycemic excursions | 72 h pre-exercise and 72 h post-exercise respectively
Heart rate variability | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, Professor, MD, Principal Investigator — University of Bern
Locations (1):
- Division of Endocrinology, Diabetes and Clinical Nutrition, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Result] Stettler C, Jenni S, Allemann S, Steiner R, Hoppeler H, Trepp R, Christ ER, Zwahlen M, Diem P. Exercise capacity in subjects with type 1 diabetes mellitus in eu- and hyperglycaemia. Diabetes Metab Res Rev. 2006 Jul-Aug;22(4):300-6. doi: 10.1002/dmrr.608. PMID 16302286
- [Result] Jenni S, Oetliker C, Allemann S, Ith M, Tappy L, Wuerth S, Egger A, Boesch C, Schneiter P, Diem P, Christ E, Stettler C. Fuel metabolism during exercise in euglycaemia and hyperglycaemia in patients with type 1 diabetes mellitus--a prospective single-blinded randomised crossover trial. Diabetologia. 2008 Aug;51(8):1457-65. doi: 10.1007/s00125-008-1045-5. Epub 2008 May 30. PMID 18512043
- [Result] Bussau VA, Ferreira LD, Jones TW, Fournier PA. The 10-s maximal sprint: a novel approach to counter an exercise-mediated fall in glycemia in individuals with type 1 diabetes. Diabetes Care. 2006 Mar;29(3):601-6. doi: 10.2337/diacare.29.03.06.dc05-1764. PMID 16505513
- [Result] Bussau VA, Ferreira LD, Jones TW, Fournier PA. A 10-s sprint performed prior to moderate-intensity exercise prevents early post-exercise fall in glycaemia in individuals with type 1 diabetes. Diabetologia. 2007 Sep;50(9):1815-1818. doi: 10.1007/s00125-007-0727-8. Epub 2007 Jun 22. PMID 17583795
- [Result] Guelfi KJ, Jones TW, Fournier PA. The decline in blood glucose levels is less with intermittent high-intensity compared with moderate exercise in individuals with type 1 diabetes. Diabetes Care. 2005 Jun;28(6):1289-94. doi: 10.2337/diacare.28.6.1289. PMID 15920041
- [Result] Guelfi KJ, Ratnam N, Smythe GA, Jones TW, Fournier PA. Effect of intermittent high-intensity compared with continuous moderate exercise on glucose production and utilization in individuals with type 1 diabetes. Am J Physiol Endocrinol Metab. 2007 Mar;292(3):E865-70. doi: 10.1152/ajpendo.00533.2006. PMID 17339500
- [Result] Iscoe KE, Riddell MC. Continuous moderate-intensity exercise with or without intermittent high-intensity work: effects on acute and late glycaemia in athletes with Type 1 diabetes mellitus. Diabet Med. 2011 Jul;28(7):824-32. doi: 10.1111/j.1464-5491.2011.03274.x. PMID 21388440
- [Result] Lecoultre V, Benoit R, Carrel G, Schutz Y, Millet GP, Tappy L, Schneiter P. Fructose and glucose co-ingestion during prolonged exercise increases lactate and glucose fluxes and oxidation compared with an equimolar intake of glucose. Am J Clin Nutr. 2010 Nov;92(5):1071-9. doi: 10.3945/ajcn.2010.29566. Epub 2010 Sep 8. PMID 20826630
- [Derived] Eckstein ML, Farinha JB, McCarthy O, West DJ, Yardley JE, Bally L, Zueger T, Stettler C, Boff W, Reischak-Oliveira A, Riddell MC, Zaharieva DP, Pieber TR, Muller A, Birnbaumer P, Aziz F, Brugnara L, Haahr H, Zijlstra E, Heise T, Sourij H, Roden M, Hofmann P, Bracken RM, Pesta D, Moser O. Differences in Physiological Responses to Cardiopulmonary Exercise Testing in Adults With and Without Type 1 Diabetes: A Pooled Analysis. Diabetes Care. 2021 Jan;44(1):240-247. doi: 10.2337/dc20-1496. Epub 2020 Nov 12. PMID 33184152
- [Derived] Bally L, Zueger T, Buehler T, Dokumaci AS, Speck C, Pasi N, Ciller C, Paganini D, Feller K, Loher H, Rosset R, Wilhelm M, Tappy L, Boesch C, Stettler C. Metabolic and hormonal response to intermittent high-intensity and continuous moderate intensity exercise in individuals with type 1 diabetes: a randomised crossover study. Diabetologia. 2016 Apr;59(4):776-84. doi: 10.1007/s00125-015-3854-7. Epub 2016 Jan 6. PMID 26739816
- [Derived] Bally L, Zueger T, Pasi N, Carlos C, Paganini D, Stettler C. Accuracy of continuous glucose monitoring during differing exercise conditions. Diabetes Res Clin Pract. 2016 Feb;112:1-5. doi: 10.1016/j.diabres.2015.11.012. Epub 2015 Dec 19. PMID 26739116